CLINICAL TRIAL: NCT03086876
Title: Clinical and Cost Effectiveness of a Parent Mediated Intervention to Reduce Challenging Behaviour in Pre-schoolers With Moderate to Severe Learning Disability: a Randomised Controlled Trial
Brief Title: Evaluation of Parent Intervention for Challenging Behaviour in Children With Intellectual Disabilities (EPICC-ID)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15/162/02
Record Dates: First submitted 2017-03-16; First posted 2017-03-22 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Challenging Behaviour

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stepping Stones Triple P (Experimental): Trained practitioners will deliver Level 4 SSTP to parents in 6 weekly group sessions and will also provide 3 telephone of face to face contacts to each participant but they will not be involved in routine care for participants in either arm. Each therapist responsible for delivering SSTP will be trained in the Group Stepping Stones Training and Accreditation programme which includes three training days and a further half day accreditation workshop after 6 weeks. The group sessions not only educate but actively train the parents in skills and the individual consultations aim to facilitate independent problem solving. The learning objectives focus on maintaining behavioural change, using skills within a group learning environment, learning from peers in the group and sharing difficulties or achievements, providing support, considering if more intensive work is required, referring further if needed, talking about risk and protective factors operating within families.
  Interventions: Behavioral: Level 4 Stepping Stones Triple P (SSTP)
- Treatment as usual (TAU) (No Intervention): TAU will be available to participants in both arms of the trial. It may include a range of services such as:
  1. Health visitor services; 2. Primary care engagement and advice; 3. Potentially some version of early intervention maybe provided by either community paediatric services or Child and Adolescent Mental Health Services, although our understanding is that very little is available for children of this age. 4. Parenting advice and support sessions by carers groups or other third sector organisations.
  Parents allocated to TAU will receive a list of national and local resources and the Contact a Family guide to challenging behavior with tips and advice on social and health care supports.

INTERVENTIONS:
Behavioral: Level 4 Stepping Stones Triple P (SSTP) — Stepping Stones Triple P is a system of psychoeducational and behavioural approaches to parenting a child with LD and challenging behaviour that aims to increase parental confidence and skills so that parents are able to manage the child's behavior effectively. SSTP comprises different levels based on increasing family complexity.
  Arms: Stepping Stones Triple P

SUMMARY:
Children with intellectual disabilities are likely to present with challenging behaviour. Parent mediated interventions have shown utility in influencing child behaviour, although there is a paucity of UK research into challenging behaviour interventions in this population. NICE guidelines favour Stepping Stones Triple P (SSTP) as a challenging behaviour intervention and this trial aims to evaluate its clinical and cost effectiveness in preschool children with moderate to severe intellectual disabilities.The trial launched in 2017 at four sites across England, with the aim of recruiting 258 participants (aged 30-59 months). The Intervention Group receive nine weeks of SSTP parenting therapy (six group sessions and three individualised face to face or telephone sessions) in addition to Treatment as Usual (TAU) whilst the TAU group receive available services in each location. Both study groups undergo the study measurements at baseline and at four and twelve months. Outcome measures include parent reports and structured observations of behaviour. Service use and health related quality of life data is also being collected to carry out a cost effectiveness and utility evaluation. Findings from this study will inform policy regarding interventions for challenging behaviour in young children with moderate to severe intellectual disabilities.

DETAILED DESCRIPTION:
About 1-2% of the population have a Learning disability (LD). This is a lifelong condition characterised by an intelligence quotient (IQ) of less than 70, general developmental delay and limitations in day to day activities. Children and adults with LD are some of the most under-served groups in society, with well documented health disparities and at four times the risk of developing a mental disorder. Reports indicate that challenging behaviour, e.g. temper tantrums, aggression or self injury, occurs in as many as 40,000 young people under 18 years living in England. There is a significant evidence from research in the general population that parenting groups which support parents in developing skills to manage such behaviours in their child can be helpful. These programmes, if offered to parents early on, may reduce and even prevent serious emotional problems and possible criminality from developing in the child later in life. Cost benefits are associated with improved health and social outcomes in the young person.

The National Institute of Health and Care Excellence (NICE) guideline on behaviour that challenges reviewed all the available evidence and found very few thoroughly researched programmes specifically developed for children and young people with LD and challenging behaviour. NICE, therefore, recommended that further research should be undertaken to address the lack of evidence based interventions to reduce challenging behaviour in the population of young people with LD.

In this study, the investigators propose to evaluate a programme called level 4 Stepping Stones Triple P (SSTP) delivered by trained practitioners to groups of parents of young children aged 30-59 months with moderate to severe LD. The programme lasts for 9 weeks and has shown positive results in small trials outside the United Kingdom, indicating that it is a potentially helpful. However, it needs to be tested within the UK health system before recommendations can be made to roll it out. Level 4 SSTP helps parents understand and manage their child's behaviour and parents may benefit from peer support in a group setting. The investigators shall recruit 258 parents who will be allocated to one of two groups by chance: one will receive SSTP and treatment as usual and the other treatment as usual, a list of resources and the Contact a Family guide to challenging behaviour. Treatment as usual includes support and advice by General Practitioner's or child development teams. The investigators shall use parental reports and observations of child behaviour to examine whether SSTP reduces challenging behaviour at four (short term) and 12 (long term) months after randomisation. They will also ask other caregivers' about the child's behaviour, the child's and the parent's health related quality of life, difficulties with care, parent stress, service use and how the parent has found the intervention using both questionnaires and face to face interviews.The investigators shall interview the service managers and the therapists about their experience of hosting and delivering the intervention. Parents will also be recruited to the Parent Advisory Group to advise about various aspects of the study, e.g. materials, interview topic guides, dissemination. The researchers and clinicians have expertise in LD, child health and early intervention and have conducted several large trials with this population. The trial will last 48 months and will follow all statutory research governance requirements to ensure that it is high quality, safe and ethical.

ELIGIBILITY:
Inclusion Criteria:

* Age: Parents 18 years or over; Child aged 30-59 months at identification;
* Child has moderate to severe intellectual disability (parent reported Adaptive Behaviour Assessment System (ABAS) General Adaptive Functioning 20-69);
* Written informed consent by parent/caregiver;
* Reports of challenging behaviour over a 6-month period but no less than 2 months.

Exclusion Criteria:

* Child has mild, profound or no LD on parent reported ABAS;
* Parent/carer has insufficient English language to complete study questionnaires;
* Another sibling is taking part in the study.

Ages: 30 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 261 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Child Behaviour Check List (CBCL) | 12 months
  Children's challenging behaviour will be measured at 12 months post randomisation using the parent completed preschool Child Behaviour Checklist (CBCL)

SECONDARY OUTCOMES:
Revised Family Observation Schedule (FOS-RIII) | 12 months
  Direct observations will be carried out by masked research assistants using the Revised Family Observation Schedule (FOS-RIII) as an objective measure of challenging behaviour
Child Behaviour Checklist Caregiver-Teacher Report Forms (C-TRF) | 12 months
  Caregiver (not parent) reported child behaviour (Child Behaviour Checklist Caregiver-Teacher Report Forms; C-TRF). Most children in the sample age range will have additional care outside the parental home allowing us to have additional perspectives on the child's behaviour.
General Health Questionnaire (GHQ) | 12 months
  We will measure parent psychiatric morbidity using the General Health Questionnaire. This well established instrument will provide additional information about common psychiatric morbidity in the parent.
Questionnaire on Resources and Stress (QRS-F short form) | 12 months
  Parent stress will be measured using the Questionnaire on Resources and Stress QRS-F short form. This validated questionnaire measures stress in caregivers of chronically ill or children with LD.
Caregiving Problem Checklist-Difficult Child Behaviour | 12 months
  Frequency of behaviour severity during care-giving tasks will be measured using the Caregiving Problem Checklist-Difficult Child Behaviour. This measure assesses the frequency of difficult child behaviour when the parent is completing care-giving tasks.
Parenting Sense of Competence Scale (PSOC) | 12 months
  Satisfaction and efficacy as parent will be measured using the Parenting Sense of Competence Scale, PSOC. The Parenting Sense of Competence scale measures parent rated competence on the dimensions of Satisfaction and Efficacy as a parent.
Child and Adolescent Service Use Schedule (CA-SUS) | 12 months
  Health and social care service use will be measured using the Child and Adolescent Service Use Schedule, CA-SUS. A modified version of the Child and Adolescent Service Use Schedule will be used in the trial.
Pediatric Quality of Life (PedsQL) | 12 months
  Health related quality of life will be measured using the Pediatric Quality of Life, PedsQL. The measure covers Physical, Emotional, Social, School Functioning domains. It contains a parent proxy report for children aged 2 years and over. It will be used in the study to derive QALYS for the health economic evaluation.
EuroQoL (EQ-5D) | 12 months
  Health related quality of life in the parent/other caregiver will be measured using the EQ-5D; 47. This self-completed questionnaire will capture parental and caregiver perspective on his/her health status which will be used in the economic evaluation.
Client Satisfaction Questionnaire (CSQ) | 4 months
  Parent intervention acceptability will be measured using the Client Satisfaction Questionnaire. The questionnaire will allow parents to provide feedback about the intervention by commenting on their satisfaction with and experience of the intervention, including ease of use, format and helpfulness. It has been specifically developed for research in SSTP.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Hassiotis, Principal Investigator — University College, London
Locations (4):
- United Kingdom (4):
  - Blackpool Teaching Hospitals NHS Foundation Trust, Blackpool
  - Central and North West London NHS Foundation Trust, London
  - Guy's and St Thomas NHS Foundation Trust, London
  - Northumberland, Tyne and Wear NHS Foundation Trust, Newcastle

REFERENCES:
- [Derived] Ondruskova T, Oulton K, Royston R; EPICC-ID Research Group; Hassiotis A. Process evaluation of a parenting intervention for pre-schoolers with intellectual disabilities who display behaviours that challenge in the UK. J Appl Res Intellect Disabil. 2024 Sep;37(5):e13263. doi: 10.1111/jar.13263. PMID 39045819
- [Derived] Ondruskova T, Royston R, Absoud M, Ambler G, Qu C, Barnes J, Hunter R, Panca M, Kyriakopoulos M, Oulton K, Paliokosta E, Sharma AN, Slonims V, Summerson U, Sutcliffe A, Thomas M, Dhandapani B, Leonard H, Hassiotis A. Clinical and cost-effectiveness of an adapted intervention for preschoolers with moderate to severe intellectual disabilities displaying behaviours that challenge: the EPICC-ID RCT. Health Technol Assess. 2024 Jan;28(6):1-94. doi: 10.3310/JKTY6144. PMID 38329108
- [Derived] Farris O, Royston R, Absoud M, Ambler G, Barnes J, Hunter R, Kyriakopoulos M, Oulton K, Paliokosta E, Panca M, Paulauskaite L, Poppe M, Ricciardi F, Sharma A, Slonims V, Summerson U, Sutcliffe A, Thomas M, Hassiotis A. Clinical and cost effectiveness of a parent mediated intervention to reduce challenging behaviour in pre-schoolers with moderate to severe intellectual disability (EPICC-ID) study protocol: a multi-centre, parallel-group randomised controlled trial. BMC Psychiatry. 2020 Jan 30;20(1):35. doi: 10.1186/s12888-020-2451-6. PMID 32000729